CLINICAL TRIAL: NCT02908399
Title: Thermal Images on Smartphones to Diagnose Bacterial Pneumonia in Children in Pakistan
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Massachusetts General Hospital (Other)
Collaborators: United States Agency for International Development (USAID) (U.S. Federal Agency)
Responsible Party: Principal Investigator, Patricia L. Hibberd, Chief, Division of Global Health, Department of Pediatrics, Massachusetts General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2016P000898
Record Dates: First submitted 2016-09-08; First posted 2016-09-21 (Estimated); Last update posted 2017-08-29 (Actual); Status verified 2017-08

CONDITIONS: Infections - Bacterial; Pneumonia - Bacterial
MeSH Terms: conditions — Bacterial Infections; Pneumonia, Bacterial

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Thermal Imaging (Experimental): Imaging using a thermal camera
  Interventions: Device: FLIR ONE

INTERVENTIONS:
Device: FLIR ONE

SUMMARY:
This is a prospective study of up to 250 participants, from birth to 18 months, who have already had a chest x-ray while a patient at the National Institute of Health (NICH) in Karachi, Pakistan. Participants will include both males and females as well as all races and ethnicities. Participants will have thermal pictures of their chest taken by trained study staff using a Smartphone and a FLIR ONE attachment. Thermal images will be read by trained radiologists to determine if bacterial pneumonia is present. Results of the thermal image will then be compared to the results of the chest x-ray. If additional images of the chest or other areas of suspected related infection are available, additional thermal images will be taken of the same location within 24 hours of the other image.

ELIGIBILITY:
Inclusion Criteria:

* 18 months or younger;
* patient at NICH Hospital in Karachi, Pakistan;
* had chest x-ray within last 24 hours to determine diagnosis of bacterial pneumonia;
* consent obtained from one parent

Exclusion Criteria:

* thermal image cannot be done within 24 hours of chest x-ray

Max Age: 18 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 250 (Estimated)
Dates: Start 2016-10; Primary Completion 2017-06 (Actual); Study Completion 2018-06 (Estimated)

PRIMARY OUTCOMES:
diagnosis of bacterial pneumonia | 24 hours
  Pneumonia is defined as the presence of an airspace opacity, lobar consolidation, or interstitial opacities on a chest x-ray. This determination will be made by two independent radiologists blinded to each other's readings, clinical information and thermal images. If they agree that pneumonia is either present or absent, that will be the final diagnosis. If there is disagreement, a third independent, blinded radiologist will break the tie.

SECONDARY OUTCOMES:
diagnosis of additional site of infection possibly related to bacterial pneumonia | up to a maximum of 28 days after original chest x-ray to diagnose pneumonia is taken
  Thermal imaging will be used to image other potential sites of infection suspected of being related to the bacterial pneumonia if suspected by physician

CONTACTS AND LOCATIONS:
Overall Officials: Patricia L Hibberd, MD, PhD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- National Institute of Child Health, Karachi, Pakistan

IPD SHARING:
Plan to Share IPD: Undecided